CLINICAL TRIAL: NCT06466954
Title: Correlation Between Spinopelvic Alignment and Uterine Dimensions in Primary Dysmenorrhea
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Randa Gomaa, Assistant Lecturer, Cairo University
Other Study IDs: P.T.REC/012/003235
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Primary Dysmenorrhea
Keywords: Spinal alignment; Pelvic alignment; Uterine dimensions; Primary Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group of Primary Dysmenorrhea: Females with Primary Dysmenorrhea
  Interventions: Other: Evaluating spinopelvic alignment parameters; Other: Measuring uterine dimensions
- Group Without Primary Dysmenorrhea: Females without Primary Dysmenorrhea
  Interventions: Other: Evaluating spinopelvic alignment parameters; Other: Measuring uterine dimensions

INTERVENTIONS:
Other: Evaluating spinopelvic alignment parameters — Evaluation of thoracic kyphosis, lumbar lordosis, pelvic tilt, and pelvic torsion
Other: Measuring uterine dimensions — Measurement of corpus length, corpus width, cervix length, and cervix width

SUMMARY:
This study was conducted to investigate the correlation between spinopelvic alignment and uterine dimensions in primary dysmenorrhea.

DETAILED DESCRIPTION:
Primary dysmenorrhea (PD) is a common condition characterized by severe menstrual cramps and lower abdominal pain before or during menstruation, without any underlying pelvic pathology. It is highly prevalent among adolescents and young women, with 16% to 93% of adolescents and 70% to 90% of young women experiencing PD. The severe menstrual discomfort associated with PD often leads to absenteeism from school or work, with approximately one-third to half of individuals missing at least one day per menstrual cycle, and 5% to 14% experiencing more frequent absences.

While the exact etiology of PD is not fully understood, researchers have proposed a potential relationship between PD and musculoskeletal factors. One hypothesis suggests that abnormal pelvic and lumbar spine alignment, coupled with abdominal muscle spasms, may affect the positioning of the uterus, increasing the susceptibility to dysmenorrhea. Additionally, lumbar spine misalignment could potentially impact uterine blood supply through vasoconstriction, contributing to menstrual pain.

Spinal misalignment has been proposed as a possible underlying cause of PD, with some studies suggesting that manual therapy techniques may alleviate PD symptoms. Furthermore, a lack of coordination between the pelvic floor muscles and surrounding soft tissues has also been implicated as a potential causative factor. However, research investigating the relationship between PD and musculoskeletal factors remains limited, and further exploration of the biomechanical factors influencing the pelvic region is needed. Therefore, this study aimed to investigate the correlation between spinopelvic alignment and uterine dimensions in primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Virginal and non-smokers.
* They should have regular menstrual cycles, verified through a three-month calendar record, with cycle durations averaging between 28 to 35 days.
* The body mass index (BMI) varied between 18.5 to 25 kg/m2.
* Additionally, girls in the study group should have moderate to severe PD (WaLIDD score ≥ 5).

Exclusion Criteria:

* Pelvic or gynecological disorders.
* Musculoskeletal disorders as low back pain.
* Spinal deformities as kyphosis and scoliosis.
* History of lower limb injuries.
* Diabetes.
* Cardiopulmonary diseases.
* Any physical impairment.
* They didn't use analgesics, non-steroidal anti-inflammatory drugs or oral contraceptives.

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: A sample of 40 girls was recruited from undergraduate students at Faculty of Physical Therapy, Cairo University and actively participated in this research.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Kyphotic angle | It was measured during the 2nd or 3rd days of menstruation for each participant in both groups.
  It was measured by a 4D formetric device as the maximum degree of kyphotic curvature, specifically the angle formed between the upper inflection point adjacent to the vertebral prominence and the thoracic-lumbar inflection point.
Lordotic angle | It was measured during the 2nd or 3rd days of menstruation for each participant in both groups.
  It was measured by a 4D formetric device as the maximum lordotic angle, calculated as the angle formed between the surface tangents at the thoracic-lumbar inflection point and the lower lumbar-sacral inflection point.
Pelvic tilt | It was measured during the 2nd or 3rd days of menstruation for each participant in both groups.
  It was determined by a 4D formetric device as the vertical disparity in millimeters (mm) between the two lumbar dimples. A positive value signifies that the right dimple is positioned higher than the left, while a negative value indicates the reverse, all in relation to a horizontal reference line connecting both dimples within the measuring system.
Pelvic torsion | It was measured during the 2nd or 3rd days of menstruation for each participant in both groups.
  It was measured by a 4D formetric device within the frontal plane, this measurement represents the degree of rotation of the right sacral dimple relative to the left sacral dimple.
corpus length | It was measured during the 2nd or 3rd days of menstruation for each participant in both groups.
  It was measured by ultrasonography. The longitudinal axis of the uterine corpus was determined at a longitudinal plane where the internal cervical os and endometrium appeared at their tallest, measured from the projection point of the endometrium on the uterine corpus to the internal cervical os.
corpus width | It was measured during the 2nd or 3rd days of menstruation for each participant in both groups.
  It was measured by ultrasonography. The transverse axis of the uterine corpus was assessed at the same plane, positioned perpendicular to the longitudinal diameter of the uterine corpus where it exhibited its maximum width.
cervix length | It was measured during the 2nd or 3rd days of menstruation for each participant in both groups.
  It was measured by ultrasonography. t was measured as the distance between the internal cervical os and the external os.
cervix width | It was measured during the 2nd or 3rd days of menstruation for each participant in both groups.
  It was measured by ultrasonography. The measurement of the transverse diameter of the uterine cervix was conducted at its thickest section, oriented perpendicular to an imaginary line corresponding to the longitudinal measurement of the cervix.

CONTACTS AND LOCATIONS:
Overall Officials: Amel M. Yousef, Prof., Study Chair — Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Cairo University, Giza, Egypt